CLINICAL TRIAL: NCT05418491
Title: A Post-intervention Follow-up of the Allergy Reduction Trial, to Investigate the Prolonged Risk Reducing Effect of a Partially Hydrolysed Infant Formula During the First Six Months of Life on Allergic Manifestations Up to the Age of 5 Years
Brief Title: The Prolonged Effect of Consumption of a Partially Hydrolyzed Infant Formula During the First 6 Months of Life on the Development of Allergic Manifestations At 5 Years of Age
Status: Completed | Type: Observational
Sponsor: FrieslandCampina (Industry)
Responsible Party: Sponsor
Other Study IDs: A.R.T. Follow-Up
Record Dates: First submitted 2022-06-10; First posted 2022-06-14 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-11

CONDITIONS: Allergy
Keywords: post-intervention, allergic manifestations
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Partially hydrolyzed protein Infant formula: Originating from A.R.T. cohort.
  Interventions: Other: No intervention is used in the current study. Interventions were given in the original A.R.T. study
- Standard infant formula: Originating from A.R.T. cohort.
  Interventions: Other: No intervention is used in the current study. Interventions were given in the original A.R.T. study
- Exclusively breastfed infants: Originating from A.R.T. cohort.
  Interventions: Other: No intervention is used in the current study. Interventions were given in the original A.R.T. study

INTERVENTIONS:
Other: No intervention is used in the current study. Interventions were given in the original A.R.T. study — The current study is a post-intervention study; interventions were given in the original A.R.T. study

SUMMARY:
The present study is a 5-year follow-up of the Allergy Reduction Trial (A.R.T.) birth cohort study of 551 infants at high-risk for allergy. The A.R.T. 5-year follow-up study, aims to investigate the prolonged effect of each feeding regimen [formula-fed (exclusively or partially) with the partially hydrolyzed formula (pHF) or the standard formula (SF), or exclusively breastfed] within the first 6 months of life on the development of any allergic manifestations up to the age of 5 years. Allergic manifestations within this time period will include the presence of any of the following: atopic dermatitis, food allergies, respiratory allergies, urticaria, drug allergy and insect venom allergy. In addition, differences on growth (weight, height, BMI) will be examined.

DETAILED DESCRIPTION:
The present study is a 5-year follow-up of the Allergy Reduction Trial (A.R.T.) birth cohort study of 551 infants at high-risk for allergy. The A.R.T. 5-year follow-up study, aims to investigate the prolonged effect of each feeding regimen [formula-fed (exclusively or partially) with the partially hydrolyzed formula (pHF) or the standard formula (SF), or exclusively breastfed] within the first 6 months of life on the development of any allergic manifestations up to the age of 5 years. Allergic manifestations within this time period will include the presence of any of the following: atopic dermatitis, food allergies, respiratory allergies, urticaria, drug allergy and insect venom allergy. In addition, differences on growth (weight, height, BMI) will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Children who were part of the Intention-to-Treat population of the A.R.T. study
* Children of the A.R.T. study ITT population within the age range of 5 years up to 5 years and 3 months
* Children of the A.R.T. study ITT population in whom at least one parent and/or legal guardian signed the written consent form

Exclusion Criteria:

* Children who did not participate in the A.R.T. study or who were not assigned to any of the 3 study arms
* Children of the A.R.T. study who are younger than 5 years of age or older than 5 years and 3 months of age
* Children of the A.R.T. study in whom parents and/or guardians do not agree to provide a written consent form

Ages: 5 Years to 63 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The target population of the present study are all the A.R.T. subjects who consisted the Intention-to-Treat (ITT) population (N=551).
Sampling Method: Non-Probability Sample
Enrollment: 455 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of allergic Manifestations | At 5 years of age
  Incidence of allergic manifestations (AM) based on parental reporting using Childhood Allergy questionnaire comparing partially hydrolyzed protein formula, standard formula and exclusive breastfeeding.

CONTACTS AND LOCATIONS:
Overall Officials: Yannis Manios, Dr., Principal Investigator — Harokopio University
Locations (3):
- Medical University of Varna, Varna, Bulgaria
- Asthma and Allergy Centre LTD, Limassol, Cyprus
- Harokopio University, Athens, Greece

IPD SHARING:
Plan to Share IPD: No